CLINICAL TRIAL: NCT04257136
Title: VBI-S for the Treatment of Hypotension in Hypovolemic Septic Shock Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Vivacelle Bio (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VBI-S-01
Record Dates: First submitted 2020-02-03; First posted 2020-02-05 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Septic Shock; Sepsis; Hypovolemia
MeSH Terms: conditions — Shock, Septic; Sepsis; Hypovolemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Treatment with VBI-S
  Interventions: Drug: VBI-S

INTERVENTIONS:
Drug: VBI-S — VBI-S is made of small particles of specific lipid called micelles and liposomes for the treatment of hypotension.

SUMMARY:
This study is being conducted to evaluate the safety and effectiveness of VBI-S in elevating the blood pressure of septic shock patients with absolute or relative hypovolemia.

DETAILED DESCRIPTION:
PURPOSE OF THE STUDY This study is being conducted to evaluate the safety and effectiveness of VBI-S in elevating the blood pressure of septic shock patients with absolute or relative hypovolemia.

STUDY TREATMENT Sepsis is a serious condition resulting from the presence of harmful microorganisms in the blood or other tissues and the body's response to their presence, leading to the malfunctioning of various organs. When hypotension due to sepsis cannot be reversed with the infusion of fluids the patient is in a state of septic shock. Septic shock is therefore an acute medical emergency and delayed therapy can lead to organ injury. VBI-S is intended to raise blood pressure in patients with septic shock.

Randomization and blinding: This is an open label study, randomization and blinding are not applicable to this study. All patients entering this study will be treated with VBI-S.

Data Safety Monitoring Board: A Data Safety Monitoring Board (DSMB) will review the study data.

Analysis Populations: * Safety Analysis Set (SAF): all patients who have received any amount of VBI-S. * Intent to treat (ITT) population: all patients who have received any amount of VBI-S

ELIGIBILITY:
Inclusion criteria:

1. Male or female at least 18 years of age
2. Evidence of bacterial infection demonstrated by positive blood culture and/or a known source of infection or an elevated procalcitonin of ≥ 2 ng/ml.
3. Patient has a mean blood pressure < 65 mmHg that is unresponsive to fluids currently available on the market.
4. Sequential Organ Failure Assessment (SOFA) score >= 5.
5. Sepsis diagnosis: The presence of infection which can be proven or suspected by 2 or more of the following criteria:

   * Lactate > 2 mmol/L
   * Mottled skin
   * Decreased capillary refill of nail beds or skin
   * Fever > 38.3˚C, or 101˚F
   * Hypothermia < 36˚C core temperature (<96.8˚F)
   * Heart rate > 90
   * Tachypnea
   * Change in mental status
   * Significant edema or positive fluid balance (>20 mL/kg over 24 hours)
   * Hyperglycemia (>140 mg/dL) in someone without diabetes
   * White blood cell count >12,000 or less than 4,000, or with >10% "bands" (immature
   * forms)
   * Elevated C-reactive protein in serum (according to your lab's cutoffs)
   * Elevated procalcitonin in serum (≥ 2 ng/ml)
   * Arterial hypoxemia (PaO2/FiO2 < 300)
   * Acute drop in urine output (<0.5 ml/kg/hr for at least 2 hours despite fluid resuscitation, or about 30 ml/hour for a 70 kg person)
   * Creatinine increase > 0.5 mg/dL
   * INR > 1.5 or aPTT > 60 seconds
   * Absent bowel sounds (ileus)
   * High bilirubin (total bilirubin > 4 mg/dL

Exclusion Criteria:

1. Patients with a ventricular assist device
2. Acute coronary syndrome
3. Pregnant
4. Bronchospasm
5. Mesenteric ischemia
6. Emergency surgery
7. Acute liver disease (Hepatitis B and C as examples)
8. Liver failure with a Model for End-Stage Liver Disease (MELD) score ≥ 19
9. Hematologic or coagulation disorders including thrombocytopenia (platelet count <50,000) and associated with hemodynamically significant active bleeding.
10. Absolute neutrophil count of < 1000 mm3
11. Current participation or participation in another experimental or device study within the last 30 days before the start of this study. Patient may be included if on other drugs for COVID-19 and or septic shock
12. Patients with a known allergy to soybeans or eggs
13. Patient is hypervolemic as assessed by CVP, ultrasound, Swan Ganz catheter, Flo-Trac, esophageal doppler, bioimpedance, ECHO, Partial carbon dioxide rebreathing (NICO), lithium dilution (LIDCO) or other method published in a peer reviewed journal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-02-17 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint of this study is the proportion of patients in whom mean blood pressure increased by at least 10 mmHg with a mean blood pressure target of 60 - 65 mmHg. | 10 Months
  The primary endpoint of this study is the proportion of patients in whom mean blood pressure increased by at least 10 mmHg with a mean blood pressure target of 60 - 65 mmHg.

SECONDARY OUTCOMES:
The secondary endpoint of this study is the proportion of patients in whom the dose of pressor drugs could be decreased after infusion of VBI-S to maintain a mean arterial pressure of 60-65 mmHg | 10 Months
  The secondary endpoint of this study is the proportion of patients in whom the dose of pressor drugs could be decreased after infusion of VBI-S to maintain a mean arterial pressure of 60-65 mmHg

CONTACTS AND LOCATIONS:
Overall Officials: Cuthbert Simpkins, MD, FACS, Principal Investigator — Vivacelle Bio
Locations (8):
- United States (8):
  - Dignity Health, Chandler, Arizona
  - University of Arizona, Tucson, Arizona
  - UMD Shock Trauma, Baltimore, Maryland
  - Adventist Health Care, Silver Spring, Maryland
  - Henry Ford Health System, Detroit, Michigan
  - Truman Medical Center, Kansas City, Missouri
  - Mount Sinai Hospital, New York, New York
  - Einstine Medical Center, East Norriton, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Simpkins C, Moncure M, Klepacz H, Roach K, Benzaquen S, Diaz-Caballero L, Cohen J, Haase D, Kumar M, DeShield H, Manasia A, Rodriguez J, Anamthathmakula P, Hurt N, Mukherjee B, Talluri K. Efficacy and safety of phospholipid nanoparticles (VBI-S) in reversing intractable hypotension in patients with septic shock: a multicentre, open-label, repeated measures, phase 2a clinical pilot trial. EClinicalMedicine. 2024 Jan 29;68:102430. doi: 10.1016/j.eclinm.2024.102430. eCollection 2024 Feb. PMID 38545092